CLINICAL TRIAL: NCT00644527
Title: "Rezeptive Musiktherapie Bei Depression - Eine Randomisierte, Placebokontrollierte Studie" / Receptive Music Therapy in Depression: A Randomized Placebo-Controlled Trial
Brief Title: Receptive Music Therapy for the Treatment of Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Vera Brandes, Paracelsus Medizinische Privatuniversität, Forschungsprogramm MusikMedizin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MIPH-2008-MT-1
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2008-11-18 (Estimated); Status verified 2008-11

CONDITIONS: Depression
Keywords: depression; music; sound; randomized controlled trial
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Listening to one of two different specific music programs (Group A), which is composed for the treatment of depressive symptoms. The music is listened to during a period of 30 minutes in the morning and 30 minutes in the evening over 5 - 15 weeks.
  Interventions: Other: Purpose designed music and sound listening program
- 2 (Experimental): Listening to one of two different specific music programs (Group B), which is composed for the treatment of depressive symptoms. The music is listened to during a period of 30 minutes in the morning and 30 minutes in the evening over 5 - 15 weeks.
  Interventions: Other: Purpose designed music and sound listening program
- 3 (Sham Comparator): Control I (Group C) : Listening 30 min in the morning and 30 min in the evening to unspecific music (Mozart) over 5 weeks.
  Interventions: Other: Sham music for depression
- 4 (No Intervention): Control II (Group D): Waiting list. - Each 50% of the subjects will be assigned randomly to either Group A (arm 1) and B (arm 2) after 5 weeks of waiting time.

INTERVENTIONS:
Other: Purpose designed music and sound listening program — Listening to one of two different specific music programs (Group A and B), which is composed for the treatment of depressive symptoms. The music is listened to during a period of 30 minutes in the morning and 30 minutes in the evening over 5 - 15 weeks.
  Other Names: Receptive Sound and Music
  Arms: 1; 2
Other: Sham music for depression — Listening 30 min in the morning and 30 min in the evening to selection of Mozart compositions over 5 weeks.
  Other Names: Mozart
  Arms: 3

SUMMARY:
Depressive symptoms are highly prevalent in the population. According to data from a Zurich longitudinal study, the lifetime incidence rate for severe depressive symptoms is 95%. Not all persons with depressive symptoms, however, need psychotherapeutic, psychiatric or pharmaceutical treatment. Many people specifically or unspecifically use music to influence their mood and clinical evidence demonstrates that active involvement in music supports an individual's treatment success during psychiatric therapy. The gray area of depressive symptoms that do not require medical treatment, but which contribute to a considerable disturbance of an individual's quality of life and ability to work, is the focus of the proposed study.

The study investigates whether listening to specific music programs arranged to influence depressive symptoms for 30 minutes in the morning and 30 minutes in the evenings can result in improvement of an individual's symptoms, as compared to listening to no prescribed music or no music treatment at all. Of specific interest is the use of music in the evening, which may contribute to the achievement of restive sleep.

The study's objective is to determine if the utilization of two specific music therapies to treat depressive symptoms, compared to a waiting list control intervention and an intervention listening to Mozart over a 5 week period, leads to an improvement of the depressive pathology among patients with moderate depressive disorders or patients with dysthymia. The study is designed as a simple blinded placebo-controlled study.

DETAILED DESCRIPTION:
Participants of this study will be recruited through radio and television programs on the topic of depressive symptomatology. The investigators assume that those who are undergoing a cycle of change between a stronger depressive mood and brightened spirits will be more likely to volunteer for study participation than those who are experiencing a period of stronger depressive mood. Consequently, we anticipate an improvement in depressive mood over the study period, even without therapy, for all participants as compared to study entry. To account for this effect, two control groups are included in the study design.

Although the anticipated effect size attributable to the specific music is relatively small, depressive symptoms are highly prevalent in the population. Therefore, from a public health perspective, even a small effect on depressive symptomology could make an important contribution to this problem as interventions could be easily designed to be applied in broad circles of the population. Furthermore, the use of specific music may be found to play a role in the future primary prevention of depressive symptoms in the population.

Sample size calculation based on on Cohen's d = 0.45. Total target for recruitment = 200 participants.

Potential participants will be targeted through advertisements on the radio and television. An internet website will be given during the radio or television advertisement. The website will only contain information about the study and an invitation to participate. Potential participants will be asked to apply by e-mail. The first 500 respondents will be sent a questionnaire in written form. Based on the estimated response rate and inclusion criteria, it is anticipated that 300 invitations for diagnostic interviews will be sent out in response to the received, completed questionnaires after the data has been imported and analyzed. From these 300 invitations, it is estimated that 200 individuals will agree to participation and will be further assessed as meeting the inclusion criteria. These 200 participants will be randomized to the intervention groups (n =100) and both control groups (n = 50 each).

Once enrolled in the study, participants will complete an advanced psychometric classification through the use of:

* BDI Beck Depression Inventory (Version II),
* HADS-D Hospital Anxiety and Depression Scale
* SCL-90-R Symptom-Checklist by L.R. Derogatis
* STAXI State-Trait Anger Expression Inventory
* STAI-G X1 abd X2 State-Trait Anxiety Inventory
* TAS-20 Toronto-Alexithymia-Scale
* PSQI Pittsburgh Sleep Quality Index
* ME Morningness/Eveningness Questionnaire (Horne and Ostberg)
* Physiological measurements: heart rate variability measurements

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 70 years with a Goldberg Depression Test Score of 15 to 65

Exclusion Criteria:

* Patients, who abuse alcohol
* Patients, with diseases as a consequence of alcohol abuse
* Patients under psychiatric treatment because of psychoses
* Patients with a Goldberg Depression Test Score of < 15 or > 65.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2008-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Change of a composite measure including the Hamilton Depression Scale (double weighted), the Beck Depression Inventory (single weighted) and the HADS-D-scale (single weighted) between study entry and 5 / 10 and 15-week-follow-up. | 15 weeks

SECONDARY OUTCOMES:
Quality of life (SF 36), Vital Exhaustion Brief Questionnaire, Primary outcome measure at 5 and 10 weeks. | 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vera Brandes, Principal Investigator — Paracelsus Medizinische Privatunsiversität, Salzburg; Joachim E Fischer, Prof MD MSc, Study Director — Mannheim Insitute of Public Health, Mannheim Medical Faculty, Heidelberg University
Locations (1):
- Psychocardiology, 2. Med. Dep., Hanusch-Krankenhaus, Heinrich Collin-Str. 30, Vienna, Austria

REFERENCES:
- [Derived] Brandes V, Terris DD, Fischer C, Loerbroks A, Jarczok MN, Ottowitz G, Titscher G, Fischer JE, Thayer JF. Receptive music therapy for the treatment of depression: a proof-of-concept study and prospective controlled clinical trial of efficacy. Psychother Psychosom. 2010;79(5):321-2. doi: 10.1159/000319529. Epub 2010 Aug 2. No abstract available. PMID 20689350